CLINICAL TRIAL: NCT01761851
Title: Metabolic and Nutritional Assessment in Patients on the Waiting List for Liver Transplantation
Brief Title: Resting Energy Expenditure in Patients on the Waiting List for Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Principal investigator, Federal University of Minas Gerais
Other Study IDs: CDS - APQ-04415-10; CDS - APQ-04415-10 (Other Grant/Funding Number: Fapemig CDS - APQ-04415-10)
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Liver Disease; Cirrhosis
Keywords: Resting metabolic rate; nutrition status; dietary intake
MeSH Terms: conditions — Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cases: Liver cirrhosis

SUMMARY:
Metabolic disorders and malnutrition are well known and have been reported in patients with chronic liver disease, but the relationship of energy metabolism and changes in nutritional status in patients on the waiting list for liver transplantation are unexplored. The aim of this study was to assess the resting energy expenditure (REE) of these patients, identifying the prevalence of hyper and hypometabolism. In addition, to assess if, malnutrition and clinical variables were associated with REE and metabolic disorders.

DETAILED DESCRIPTION:
This cross-sectional and descriptive study was carried out at the Alfa Institute of Gastroenterology, Hospital of Clinics, Universidade Federal of Minas Gerais (UFMG). The research protocol was approved by the UFMG Ethics Committee. Patients with indication for liver transplantation, aged over 20 years who regularly attended the Liver Outpatient Transplant Clinic were included after having agreed and signed the informed consent form. The presence of endocrine abnormalities (hyper/hypothyroidism) and patients on the waiting list for a double or re-transplant were excluding conditions. The REE and nutritional status assessment were performed by the same trained investigator (LGF) in order to reduce errors.

Resting Energy Expenditure - REE was measured by indirect calorimetry using a gas analyzer K4b2 (Cosmed, Rome, Italy). The test was performed in a silent, temperature-controlled room (22-24oC) in the morning, between 08:00am and 09:30am. The patients fasted for 12 hours, and remained on the lying position for about 20 minutes before the beginning of the test. The device was calibrated before each exam. The volume of inspired oxygen (VO2) and exhaled carbon dioxide (VCO2) was collected through a turbine and a sample line, adapted to the face mask, applied to the patient and, connected to the unit. The collection of gases occurred for 25 minutes, and the first 5 minutes were discarded. The mean VO2 and VCO2 per minute were used to calculate the REE according to the Weir formula. The obtained data were multiplied by 1,440 to obtain the 24-hour REE. Therefore, the REE was divided by kilograms of fat free mass - FFM (REE/FFM). Predicted REE was calculated from the Harris and Benedict formula (REEHB). In patients with fluid retention (clinical evidence of ascites and/or limb edema) dry weight was calculated by deducting an estimated weight for ascites and/or limb edema. Hypermetabolic patients were identified if the ratio REE:REEHB was > 120% and hypometabolic patients were classified according to the ratio REE:REEHB < 80%. The non-protein respiratory quotient (RQ) was calculated by the formula VCO2/VO2. Oxidation rates of carbohydrate and fat were expressed as percentages of total generated energy.

Nutritional Assessment - Nutritional status was provided by the Subjective Global Assessment (SGA), anthropometric measurements, handgrip strength, bioimpedance and energy balance (EB) analyses. The SGA adapted for patients on the waiting list for liver transplantation is based on clinical history and physical examination, as well as the presence of existing conditions such as encephalopathy, chronic or recurrent infection, varicose veins and renal function. Patients were classified as nourished and those classified as suspected or moderately malnourished and severely malnourished were grouped together to form the malnourished group.

Anthropometric evaluation was comprised of weight, height, body mass index (BMI), triceps and subscapular skinfold thickness (TSF and SSF respectively, measured with the Lange Skinfold Caliper - Cambridge Scientific Industries Inc., Cambridge, MD, USA), midarm circumference (MAC, measured with inextensible tape), arm muscle area (AMA) and arm fat area (AFA). To minimize practical variability, the average of three consecutive measurements was recorded. Values of TSF, SSF, MAC, AMA and AFA below the 5th percentile and BMI below 18.5kg/m2 (or 22.0kg/m2 for elderly) were considered as malnutrition.

Handgrip strength (HS) was assessed with the Jamar Handgrip Dynamometer (Preston, Jackson, MI, USA) using the non-dominant arm, and the mean of three measurements was determined. Malnutrition was defined as values of HS below the 5th percentile.

Bioelectrical impedance analysis (Quantum X - RJL Systems, Inc., Clinton Township, Michigan) was used to determine body composition. Measurements were made with patients lying in bed with 4 electrodes attached to the dorsum of the right hand and foot. Phase angle (PA), fat mass (FM - kg), fat free mass (FFM, kg), total body water (TBW - L), intracellular water (ICW - L) and extracellular water (ECW - L), were evaluated. PA was categorized in equal to or less than 5.4o, or above 5.4o as proposed by Selberg et al.

The energy balance (EB) was obtained by subtracting the total energy expenditure from the total caloric intake (TCI). The TEE was obtained by multiplying the 24-hour REE by the calculated activity factor (AF), which was based on the description of the patients' daily activities and the corresponding computed values of metabolic equivalents (METs). Food intake was assessed by a 3-day food record (DietPro5i® Agromídia Software, Viçosa, Brazil).

Clinical and other variables - Age, sex, etiology, severity of liver disease by the Child-Pugh score (22) and the Model for End Stage Liver Disease score (MELD), complications like presence of fluid retention and hepatic encephalopathy; number of medication and diuretics; β-blockers and lactulose use were all compiled. Diagnosis of liver cirrhosis was based of clinical, biochemical and histopathological data. The indications for liver transplantation were categorized into alcoholic cirrhosis, viral and other diseases. Liver function tests (aspartate aminotransferase - AST, alanine aminotransferase- ALT, total bilirubin-TB and international normalized ratio-INR), presence of diabetes and/or glucose intolerance (24) and fasting glucose were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* all patients who agreed to participate and signed the informed consent

Exclusion Criteria:

* those who refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the waiting list for liver transplant
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | 12 months
  Assess resting energy expenditure

SECONDARY OUTCOMES:
Metabolic alterations - hyper or hypo metabolism | 12 months
  Assess the metabolic status of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Maria Isabel TD Correia, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Ambulatório de Transplantes Hepáticos, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Montejo Gonzalez JC, Mesejo A, Bonet Saris A; Metabolism and Nutrition Working Group of the Spanish Society of Intensive Care Medicine and Coronary units. Guidelines for specialized nutritional and metabolic support in the critically-ill patient: update. Consensus SEMICYUC-SENPE: liver failure and liver transplantation. Nutr Hosp. 2011 Nov;26 Suppl 2:27-31. doi: 10.1590/S0212-16112011000800006. PMID 22411515
- [Background] Lee WG, McCall JL, Gane EJ, Murphy R, Plank LD. Oral beta-blockade in relation to energy expenditure in clinically stable patients with liver cirrhosis: a double-blind randomized cross-over trial. Metabolism. 2012 Nov;61(11):1547-53. doi: 10.1016/j.metabol.2012.04.001. Epub 2012 May 4. PMID 22560128
- [Background] Anastacio LR, Ferreira LG, Ribeiro Hde S, Lima AS, Vilela EG, Correia MI. Weight loss during cirrhosis is related to the etiology of liver disease. Arq Gastroenterol. 2012 Jul-Sep;49(3):195-8. doi: 10.1590/s0004-28032012000300005. PMID 23011241
- [Background] Ferreira LG, Anastacio LR, Correia MI. The impact of nutrition on cirrhotic patients awaiting liver transplantation. Curr Opin Clin Nutr Metab Care. 2010 Sep;13(5):554-61. doi: 10.1097/MCO.0b013e32833b64d2. PMID 20531175